CLINICAL TRIAL: NCT01292837
Title: An Open-label, Single-arm, Multicenter Study to Evaluate the Efficacy and Safety of Adjunctive Treatment With Levetiracetam in Japanese Patients (≥4 to <16 Years) With Uncontrolled Generalized Tonic-clonic (GTC) Seizures Despite Treatment With 1 or 2 Antiepileptic Drug(s)
Brief Title: A Study of Levetiracetam in Japanese Pediatric Patients With Generalized Tonic-clonic Seizures
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Japan Co. Ltd. (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N01363; 2014-004382-25 (EudraCT Number)
Record Dates: First submitted 2011-02-08; First posted 2011-02-10 (Estimated); Results first posted 2014-08-12 (Estimated); Last update posted 2015-05-15 (Estimated); Status verified 2015-04

CONDITIONS: Epilepsy; Generalized Tonic-clonic Seizures
Keywords: Levetiracetam; Epilepsy; Generalized tonic-clonic seizures
MeSH Terms: conditions — Epilepsy; Seizures | interventions — Levetiracetam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Levetiracetam (Experimental): Twice daily (morning and evening) orally
  Interventions: Drug: Levetiracetam

INTERVENTIONS:
Drug: Levetiracetam — The initial dose is 20 mg/kg/day or 1000 mg/day, divided into two equal dose for the first two weeks, followed by 40 mg/kg/day or 2000 mg/day for two weeks. After reaching 60 mg/kg/day or 3000 mg/day, treatment will continue for 20 weeks.
  Other Names: Keppra; E Keppra

SUMMARY:
To evaluate the efficacy and safety of Levetiracetam dry syrup at doses up to 60 mg/kg/day or 3000 mg/day used as adjunctive therapy in Japanese pediatric patients aged ≥4 to <16 years with uncontrolled Generalized Tonic-Clonic (GTC) seizures despite treatment with 1 or 2 Anti-Epileptic Drugs (AEDs).

ELIGIBILITY:
Inclusion Criteria:

* An epileptic patient with generalized tonic-clonic seizures that are classifiable according to the International League Against Epilepsy classification of epileptic seizures (Epilepsia, 1981)
* A patient on a stable dose of 1 or 2 anti-epileptic drugs for the last 4 weeks (potassium bromide and sodium bromide for the last 12 weeks) prior to the Combined Baseline Period and during the Combined Baseline Period

Exclusion Criteria:

* Presence of any sign (clinical or imaging procedures) suggesting a progressive brain lesion/disease, in particular, progressive disorder with epileptic seizures
* Diagnosis of Lennox-Gastaut Syndrome
* Confirmed focal epilepsy based on clinical signs (seizure types), with consistent electroencephalogram and magnetic resonance imaging features
* A history of convulsive or nonconvulsive status epilepticus while taking concomitant anti-epileptic drugs for the last 3 months prior to Visit 1

Ages: 4 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 13 (Actual)
Dates: Start 2011-02; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (26):
- Japan (26):
  - 191, Akita
  - 184, Bunkyō City
  - 309, Bunkyō City
  - 107, Gifu
  - 303, Hiroshima
  - 108, Kobe
  - 302, Kodaira
  - 306, Kōshi
  - 136, Moriyama
  - 305, Nagoya
  - 190, Nerima City
  - 125, Neyagawa
  - 301, Niigata
  - 116, Ohmura
  - 109, Okayama
  - 308, Ōnojō
  - 119, Saitama
  - 117, Sapporo
  - 304, Sapporo
  - 103, Sendai
  - 138, Shimotsuke
  - 307, Shizuoka
  - 139, Takatsuki
  - 135, Tsu
  - 193, Yokohama
  - 310, Yufu

REFERENCES:
- See also: FDA safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This multicenter study started to enroll subjects in Februray 2011 in order to end up with 8 sites in Japan with enrolled subjects.
  Participant Flow refers to the Enrolled Set (ES). ES consists of all subjects who signed the consent form and participated in the Prospective Baseline Period.
Period: Overall Study
Arm/Group | Levetiracetam
Started | 13
Completed | 11
Not Completed | 2
Not completed — Adverse Event | 1
Not completed — Further treatment determined | 1

BASELINE CHARACTERISTICS:
Population: The Baseline Analysis Population refers to the Safety Set. The Safety Set was a subset of the Enrolled Set and consisted of all subjects taking at least 1 dose of the study medication.
Arm/Group | Levetiracetam
Number analyzed (Participants) | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.7 (4.1)
Age, Customized [Number; unit: participants]
  ≥4 to <8 years | 4
  ≥8 to <12 years | 2
  ≥12 to <16 years | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 9
Region of Enrollment [Number; unit: participants]
  Japan | 13
Weight [Mean (Standard Deviation); unit: kilogram] | 32.22 (16.56)
Height [Mean (Standard Deviation); unit: centimeter] | 129.36 (26.32)
Body Mass Index [Mean (Standard Deviation); unit: kilogram per squaremeter (kg/m^2)] | 17.89 (3.75)

OUTCOME MEASURES:

1. Primary Outcome: The Percent Change From the Combined Baseline (4-week Retrospective Baseline and 4-week Prospective Baseline) in the Generalized Tonic-clonic Seizure Frequency Per Week Over the 24-week Treatment Period (Up-Titration and Evaluation Periods)
Description: The percent change from Combined Baseline over Treatment Period was calculated from the Generalized Tonic-Clonic (GTC) seizure frequency per week during the Treatment Period (T) and during the Baseline Period (B, Combined Baseline, ie, Retrospective and Prospective Baseline Periods) using the equation below.
  The percent change from Baseline = (B - T)/B x 100
  The seizure frequency per week was calculated using the following formula:
  Frequency per week of GTC seizures = total number of GTC seizures in the corresponding period / number of days for observation in the corresponding period x 7
Time Frame: From Baseline (Week -8) to Treatment Period (Week 0 to Week 24)
Population: The Analysis Population refers to the Full Analysis Set (FAS). The FAS was a subset of the Safety Set and included all subjects with Combined Baseline Period (Retrospective and Prospective) and post-Baseline Generalized Tonic-Clonic seizure counts as the primary efficacy analysis.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Levetiracetam
Number analyzed (Participants) | 13
percent change | 45.47 (50.34)

2. Secondary Outcome: The Percent Change in Generalized Tonic-clonic Seizure Frequency Per Week From the Combined Baseline Period Over the Evaluation Period
Description: The percent change from Combined Baseline over Evaluation Period was calculated from the Generalized Tonic-Clonic (GTC) seizure frequency per week during the Evaluation Period (E) and during the Baseline Period (B, Combined Baseline, ie, Retrospective and Prospective Baseline Periods) using the equation below.
  The percent change from Baseline = (B - E)/B x 100
  The seizure frequency per week was calculated using the following formula:
  Frequency per week of GTC seizures = total number of GTC seizures in the corresponding period / number of days for observation in the corresponding period x 7
Time Frame: From Baseline (Week -8) to Evaluation Period (Week 4 to Week 24)
Population: The Analysis Population refers to the Full Analysis Set (FAS). The FAS was a subset of the Safety Set and included all subjects with combined Baseline Period and post-Baseline generalized tonic-clonic seizure counts. 12 of the 13 subjects in the FAS were included in the analysis excluding 1 subject discontinued before the Evaluation Period.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Levetiracetam
Number analyzed (Participants) | 12
percent change | 44.93 (51.86)

3. Secondary Outcome: Generalized Tonic-clonic Seizures 50 % Responder Rate (the Proportion of Subjects With 50 % or More Reduction From the Combined Baseline in the Frequency of Generalized Tonic-clonic Seizures) During the Treatment Period
Description: The 50 % responder rate during the Treatment Period was the proportion of subjects who reported a ≥ 50 % reduction in seizure frequency per week from Baseline during the Treatment Period.
Time Frame: From Baseline (Week -8) to Treatment Period (Week 0 to Week 24)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Levetiracetam
Number analyzed (Participants) | 13
percentage of participants | 53.8

4. Secondary Outcome: Generalized Tonic-clonic Seizures 50 % Responder Rate During the Evaluation Period
Description: The 50 % responder rate during the Evaluation Period was the proportion of subjects who reported a ≥50 % reduction in seizure frequency per week from Baseline during the Evaluation Period.
Time Frame: From Baseline (Week -8) to Evaluation Period (Week 4 to Week 24)
Population: The Analysis Population refers to the Full Analysis Set (FAS). The FAS was a subset of the Safety Set and included all subjects with Combined Baseline Period (Retrospective and Prospective) and post-Baseline Generalized Tonic-Clonic seizure counts as the primary efficacy analysis.
  One subject discontinued the study during the Up-Titration Period.
Measure: Number; unit: percentage of participants
Arm/Group | Levetiracetam
Number analyzed (Participants) | 12
percentage of participants | 58.3

5. Secondary Outcome: Generalized Tonic-clonic Seizure Freedom Over the Treatment Period
Description: A subject with a generalized tonic-clonic seizure frequency of 0 per week throughout the Treatment Period was considered a seizure-free subject for that period.
Time Frame: Treatment Period (Week 0 to Week 24)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Levetiracetam
Number analyzed (Participants) | 13
participants | 2

6. Secondary Outcome: Generalized Tonic-clonic Seizure Freedom Over the Evaluation Period
Description: A subject with a generalized tonic-clonic seizure frequency of 0 per week throughout the Evaluation Period was considered a seizure-free subject for that period.
Time Frame: Evaluation Period (Week 4 to Week 24)
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Levetiracetam
Number analyzed (Participants) | 12
participants | 2

ADVERSE EVENTS:
Time Frame: Treatment Emergent Adverse Events were reported from Baseline up to Week 30
Description: The Analysis Population refers to the Safety Set. The Safety Set was a subset of the Enrolled Set and consisted of all subjects taking at least 1 dose of the study medication.
Arm/Group | Levetiracetam
Serious Adverse Events (participants affected / at risk) | 0/13
Other Adverse Events (participants affected / at risk) | 13/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Levetiracetam (N=13)
Diarrhoea (Gastrointestinal disorders) | 2 (5)
Nasopharyngitis (Infections and infestations) | 3 (5)
Convulsion (Nervous system disorders) | 3 (5)
Somnolence (Nervous system disorders) | 3 (3)
Dental caries (Gastrointestinal disorders) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 1 (1)
Pyrexia (General disorders) | 1 (2)
Impetigo (Infections and infestations) | 1 (1)
Otitis media (Infections and infestations) | 1 (1)
Pneumonia mycoplasmal (Infections and infestations) | 1 (1)
Arthropod sting (Injury, poisoning and procedural complications) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 1 (1)
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 1 (1)
Electrocardiogram QT prolonged (Investigations) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Bradykinesia (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory tract haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
Excessive granulation tissue (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days